CLINICAL TRIAL: NCT01379612
Title: Ultrasound Elastography of Rectal Cancer Patients Treated With Preoperative Chemoradiation
Brief Title: Ultrasound Elastography in Patients With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-20100028
Record Dates: First submitted 2011-06-08; First posted 2011-06-23 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Rectal Cancer
Keywords: Ultrasound elastography; Rectal cancer; Preoperative chemoradiation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal cancer patients in chemoradiation
  Interventions: Other: Ultrasonic Elastography

INTERVENTIONS:
Other: Ultrasonic Elastography — Non-invasive

SUMMARY:
The aim of this study is to recruit 50 rectal cancer patients planned to receive standard radiochemotherapy. A baseline ultrasonic elastography is performed prior to radiochemotherapy and followed by re-scans two and six weeks after initiation of treatment. The objective quantitative elastography findings are compared with the TRG score.

The purpose is to elucidate ultrasonic elastography's ability to predict treatment response at an early stage by comparing quantitative ultrasound parameters before, during and after treatment with MR scan results and histopathological Tumor Regression Grade (TRG score) after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy verified adenocarcinoma in the rectum ≤ 10 cm from the anal verge.
2. T3/4 tumor assessed by transrectal ultrasound and MR, and CRMMR < 5 mm.
3. Life expectancy of more than 3 months.
4. Age ≥18 years.
5. Performance status ≤ 2 according to WHO.
6. Patient able to observe protocol guidelines.
7. Signed informed consent.

Exclusion Criteria:

1. Previous radiation treatment for the pelvis.
2. Known distant metastases.
3. Serious disease contraindicating treatment, including cardiovascular disease.
4. Other malignant disease apart from curativly treated non-melanotic skin cancer and previously treated carcinoma in situ cervicis uteri.
5. Pacemaker
6. other disease making the patient unfit for study participation as assessed by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients planned for preoperative chemoradiation at the Dept. of Oncology, Vejle Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tumor regression grade | 8 weeks after operation

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Dept. of Oncology, Vejle Hospital, Vejle
  - Dept. of Radiology, Vejle Hospital, Vejle